CLINICAL TRIAL: NCT01915628
Title: A Canadian Pre-market Registry of the BioMatrix Flex™ Drug Eluting Stents.
Brief Title: e-BioMatrix Canada Registry
Status: Completed | Type: Observational
Sponsor: Biosensors Europe SA (Industry)
Responsible Party: Sponsor
Other Study IDs: 11-EU-02
Record Dates: First submitted 2013-07-30; First posted 2013-08-05 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Device Related MACE and Bleeding
Keywords: MACE; Safety; Efficacy; On label; Myocardial Infarction; Cardiac death; TVR; stent thrombosis
MeSH Terms: conditions — Hemorrhage; Myocardial Infarction; Death

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BioMatrix Flex: percutaneous coronary intervention
  Interventions: Device: BioMatrix Flex

INTERVENTIONS:
Device: BioMatrix Flex — Percutaneous coronary intervention

SUMMARY:
Prospective, multi-center registry to be conducted at 6 Canadian interventional cardiology centers. The e-BioMatrix data will be compared with a historical control group, the Cypher arm of the Biosensors Leaders study consisting of 313 patients. All patients will be followed for up to 2 years.

DETAILED DESCRIPTION:
The purpose of this registry is to capture additional "on-label" clinical data of the CE-marked BioMatrix Flex™ (BA9™-Eluting) stent system in relation to safety and effectiveness.

This prospective, multi-center registry will enroll a total of 533 patients. The BioMatrix FlexTM has been studied in randomized controlled trials and has been granted the CE mark. The data have been reviewed by Health Canada and no further randomized trials were requested. Prior to marketing approval, Health Canada requested that a registry be implemented to provide data in Canada on 'on label patients' to supplement the data already available from the Leaders trial, conducted on 'all comers' patients. The registry follows the normal medical practice for drug eluting stents in Canada. 100% informed consents will be checked, and at least all Major Adverse Cardiac Events up to 2 years will be source data verified. All MACEs developing in the patient population will be adjudicated by an independent Clinical Events Committee. The patients will be followed clinically for up to 2 years after stent implantation.

A third party Contract Research Organisation, Centre for Innovative Medicine has has been appointed to perform site monitoring and project management.

The appropriate Data Management and Validation, Statistical Analysis, Safety, Monitoring Plans and guidelines have been put into place to address quality and consistency of data.

A Clinical Event Committee (CEC) has been put in place for this registry, consisting of cardiologists not participating in the registry. The mandate of this CEC will be to review all Major Adverse Cardiac Events (MACE), to adjudicate and to classify them. In addition, and in order to protect study participants, there will be a regular review of all reported safety events by the sponsor Clinical Safety Officer and a weekly assessment of the incidence of the important risks pertaining to the registry in order to detect any safety signals.

The sites have been trained during the Site Initiation Visits on registry operations and analysis activities, such as patient recruitment, data collection, data management, data analysis, reporting for adverse events, and change management.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Presence of coronary artery stenosis in one or two native coronary arteries from 2.25 to 4.0 mm in diameter that can be each covered with one BioMatrix FlexTM stent
3. Up to two lesions in two separate vessels to be treated

Exclusion Criteria:

1. Inability to provide informed consent;
2. Life expectancy less than 2 years;
3. Staged procedure planned within index procedure hospitalization;
4. ST elevation myocardial infarction;
5. Angiographic evidence of thrombus;
6. EF < 20%;
7. Coronary artery bypass graft-lesion incl SVG;
8. Chronic total occlusion of the target lesion;
9. In stent restenosis
10. Bifurcation requiring 2 or more stents;
11. Left Main lesion;
12. Renal insufficiency (serum creatinine > 260 µmolmol/L or > 2.95mg/dl)
13. Multi-vessel disease with more than two vessels affected;
14. Have known intolerance to aspirin, clopidogrel, heparin, stainless steel, Biolimus A9 (limus compounds), contrast material;
15. Currently participating in another study;
16. Planning to have surgery within 6 months (excluding surgery which DAPT is maintained throughout the peri-surgical period);
17. Woman of childbearing potential with a positive pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for percutaneous coronary intervention with lesions suitable for stent implantation will be included according to the inclusion and exclusion criteria specified below.
Sampling Method: Non-Probability Sample
Enrollment: 535 (Actual)
Dates: Start 2013-05; Primary Completion 2016-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Registry device-related MACE | 12 months
  Registry device oriented major adverse cardiac events (MACE) plus bleeding events in the overall population, defined as composite of cardiac death, myocardial infarction (Q-wave and non-Q-wave), or justified target vessel revascularization at 12 months.

SECONDARY OUTCOMES:
Primary and secondary stent thrombosis | 30days, 6 months, 12 months and 2 years
  definite and probable according to ARC definitions
Registry device oriented major adverse cardiac events (MACE) in the overall population | 30d, 6m and 2y
  Defined as composite of cardiac death, myocardial infarction (Q- wave and non-Q-wave), or justified target vessel revascularization
Individual MACE components | 30d, 6m, 12m and 2y
  cardiac death, myocardial infarction, justified target vessel revascularization and bleeding events)
Bleeding per BARC criteria | 30d, 6m, 12m, 2y;
  BARC 3 to 5, all BARC, by vascular access site (femoral/radial)
Patient Oriented Composite Endpoint | 30d, 6m, 12m, 2y
  Defined as any cause mortality, MI (Q-wave and non-Q-wave), or any clinically driven target vessel revascularization;
Death and MI | 30d, 6m, 12m, 2y
Death and post-procedural MI | 30d, 6m, 12m, 2y
Antiplatelet compliance | 30d, 6m, 12m, 2y

OTHER OUTCOMES:
Sub analyses | through 2y
  Small vessel disease; Diabetic patients; Acute coronary syndrome versus no acute coronary syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Luc Bilodeau, MD, Principal Investigator — Royal Victoria Hospital, Montreal, Canada
Locations (4):
- Canada (4):
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - Sunnybrook Health Sciences, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Royal Victoria Hospital, Montreal, Quebec